

# Official Title: Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation

Date of Protocol: September 28, 2021

NCT Number: NCT05083351





Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin **Pigmentation** 

**Revision:** 

**Clinical Investigation Title:** 

Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin

Pigmentation

Clinical Investigation Number, Version:

Other Study Identifier: N/A

Masimo MightySat<sup>TM</sup> - Investigational Study Device(s):

Optional: other FDA-cleared or commercially available pulse oximetry sensors

Sponsor: Masimo Corporation

52 Discovery

Irvine, California 92618 USA





Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin **Pigmentation** 

**Investigator Page** 

Principal Investigator (s):



Investigation Site(s): Masimo Corporation – Clinical Lab

> 52 Discovery Address: Irvine, CA 92618

> > IRB: E&I West Coast Board – IRB00007807

304 SE 3rd Street Address:

Lee's Summit, MO 64063

Agreement between Investigator and Sponsor Regarding Responsibilities for Good Clinical Practice

International Conference of Harmonization (ICH) E6 Good Clinical Practice guidance is an international ethical and scientific quality standard for designing, conducting, recording, and reporting trials that involve the participation of human subjects. It specifies general requirements intended to:

- Protect the rights, safety and well-being of human subjects,
- Ensure the scientific conduct of the clinical investigation and the credibility of the clinical investigation results,
- Assist sponsors, monitors, investigators, ethics committees, regulatory authorities and other bodies involved in the conformity assessment of medical devices.

The Principal Investigator of the clinical investigation shall:

- Obtain and maintain IRB approval of the study.
- Ensure all subjects are consented prior to enrollment, per FDA Code of Federal Regulations titled 21 CFR 50.
- Ensure only appropriately trained personnel will be involved in clinical investigation.
- Maintain study records mentioned in the Clinical Investigation Plan.
- Maintain logs for study team delegation, site visit/monitoring, equipment disposition, study team training, subject recruitment and enrollment.
- Evaluate all adverse events and adverse device effects and determining whether the study is safe to continue.
- Allow the sponsor to conduct periodic monitoring of study activities to ensure GCP compliance.
- Not promote device prior to clearance by FDA for commercial distribution, except for academic purposes and scientific presentations.

The Sponsor shall ensure existence and record of all necessary compliance documents and will conduct monitoring visits to ensure appropriate conduct of the study.

The principal investigator's signature on this page constitutes the investigator's affirmation that he or she is qualified to conduct the clinical investigation, agreement to adhere to all stipulations of this clinical investigation plan, the conditions of the Institutional Review Board (IRB) or Research Ethics Committee approval, federal and local regulatory requirements, 21 CFR 812, ISO 14155, and International Conference on Harmonization Good Clinical Practice (ICH GCP) guidance.

| Principal Investigator: | Title: | Signature: | Date: |
|-------------------------|--------|------------|-------|
| Sponsor Representative: | Title: | Signature: | Date: |





Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation

## 1. OVERALL SYNOPSIS OF THE CLINICAL INVESTIGATION

| Clinical investigation title: | Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation |
|---|---|
| Study objective(s): | The primary objective of this study is to evaluate the noninvasive oxygen saturation (SpO2) performance of the noninvasive Masimo MightySat against reference arterial blood samples analyzed by a laboratory CO-oximeter reference instrument. The study will include different subgroups to assess the performance across different genders and skin pigmentation. An optional secondary objective of this study may be to evaluate other pulse oximetry sensors for research purposes. These sensors may include other FDA-cleared devices and commercially available pulse oximeters. |
| Investigational device(s): | Masimo MightySat |
| Number of subjects: | A minimum of 36 subjects. |
| Inclusion criteria: | Refer to Section 6.3.1. |
| Exclusion criteria: | Refer to Section 6.3.1. |
| Duration of the clinical investigation: | Expected duration of study enrollment is 3 to 6 months. Subject participation in the study will be approximately 180 minutes. |
| Study endpoint(s): | Validation of the SpO2 performance of MightySat |

### 2. IDENTIFICATION AND DESCRIPTION OF THE INVESTIGATIONAL DEVICE

## 2.1. Background and Study Devices

An invasive blood sample analyzed by a CO-oximeter reference instrument gives the best measure of arterial oxygen concentration as well as other blood solutes but cannot measure these parameters continuously and requires skin puncture, arterial line placement and subsequent risk of infection, hematoma, and other physiological damage.

Masimo Corporation develops non-invasive medical technologies. These devices have applications in the operating room, critical care unit, emergency room, emergency transport vehicles, alternative (home) care, as well as physicians' offices. Masimo SET, Masimo rainbow, and other newly developed Masimo technology allow real-time, non-invasive monitoring of oxygen saturation. Use of monitoring devices on patients has the potential to improve clinical outcomes while reducing the cost of care and risks to both patients and clinicians associated with arterial and venous punctures.

The investigational MightySat used in this study is similar to the commercially available MightySat except that it has an updated SpO2 (functional oxygen saturation) calibration that was made as part of the product's continued improvements. MightySat is a stand-alone fingertip pulse oximeter that combines the functionality of a pulse oximeter monitor and sensor into a single portable device that fits on a user's finger. The device is capable of calculating SpO2 and pulse rate (PR) as well as other pulse oximeter parameters (e.g. perfusion index, respiration rate, etc.).

Other FDA-cleared or other commercially available pulse oximeters may be used for research purposes.

## 2.2. Site Information

The Masimo Clinical Laboratory facility is designed as a Phase 1 clinical study research center. The laboratory is staffed by physicians, anesthesiologists, certified registered nurse anesthetists, registered nurses, medical assistants, and clinical research staff. All personnel undergo required routine training on GCP and human research subject protections. The laboratory is equipped with standard FDA-approved medical monitoring equipment including ECG monitors, blood pressure monitors, pulse oximeters, standard hematology analyzers, and has emergency crash carts available. Hospitals and urgent care facilities are within three miles of the Masimo Clinical Laboratory.





Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation

## 3. JUSTIFICATION FOR THE DESIGN OF THE CLINICAL INVESTIGATION

This study is designed to compare the performance of the MightySat as the subjects undergo a controlled desaturation protocol. This type of study design is required to evaluate the performance of pulse oximeters based upon the ISO 80601-2-61 standard which is also adopted and referenced by the FDA.

# 4. BENEFITS AND RISKS OF THE INVESTIGATIONAL DEVICE, CLINICAL PROCEDURE, AND CLINICAL INVESTIGATION

### 4.1. Benefits:

There will be no benefit to the subject. Other possible benefits would be to society as a whole. Evaluation of the accuracy of this new device could enable users to more appropriately monitor and identify potentially life-threatening conditions.

## 4.2. Risks/Discomforts:

### • Device Risks:

The noninvasive devices used in this study are similar in technology and design to some commercially available pulse oximeters and other non-invasive devices and hence have the same risks. Pulse oximeters and other non-invasive devices are commonly used and are considered to be minimal risk.

There is an extremely small risk of damage to the subject's fingers, or other locations where sensors are placed from the device, including temporary skin irritation or discomfort associated with exposure to the sensor, as well as potential temporary mechanical irritation or discomfort. There is a remote, yet possible, risk of a burn from the sensor. In the case of a sensor burn, there is the potential for permanent skin damage (scar/discoloration).

If there are any cuts and/or abrasions near the fingernail, certain types of sensors may not be placed on that finger to avoid any discomfort for the subject.

### Venous Cannulation Risks:

Risks associated with venipuncture include discomfort, bruising, bleeding, swelling, infection, hematoma, decreased blood supply, damage to the blood vessel and surrounding nerves, tendons, or tissue, and loss of feeling in the hand and/or arm.

Other anticipated adverse events that may occur, include but are not limited to: vasovagal syncope (fainting), infiltrated IV, blood clot, lightheadedness, feeling flush/warm, feeling nauseated, throwing up, seizures, sudden drop in blood pressure/sudden increase in blood pressure, sudden drop in heart rate/sudden increase in heart rate, tingling sensation of face, arms and/or legs, sweating, and/or mouth dryness.

These anticipated adverse events are expected to be temporary.

### • Arterial Cannulation Risks:

Risks include bleeding, decreased blood supply, swelling, infection, bruising, hematoma, damage to the blood vessel and surrounding nerves, tendons, or tissue. Additional risks include vasovagal syncope (fainting), lightheadedness, feeling flush/warm, embolization (blood clot), feeling nauseated, throwing up, seizures, sudden drop in blood pressure/sudden increase in blood pressure, sudden drop in heart rate/sudden increase in heart rate, tingling sensation of face, arms, and/or legs, sweating, mouth dryness, arterial occlusion, arterial laceration, loss of feeling in the hand and/or arm, and even the loss of the hand due to rare complications of the study.

## • Blood Draw Risks:

Discomfort is generally associated with needle puncture. The most common complications associated with blood draws are hematomas or bruising. There is also a possible risk of infection, tendon or tissue damage, damage to the blood vessel and surrounding nerves, inadvertent arterial puncture, and/or loss of feeling in the hand and/or arm.





Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation

Other anticipated adverse events that may occur, include but are not limited to: vasovagal syncope (fainting), lightheadedness, feeling flush/warm, feeling nauseated, throwing up, seizures, sudden drop in blood pressure/sudden increase in blood pressure, sudden drop in heart rate/sudden increase in heart rate, tingling sensation of face, arms and/or legs, sweating, and/or mouth dryness. These anticipated adverse events are expected to be temporary.

## • Risk From Oxygen Administration:

It is expected that some people may experience feelings of claustrophobia or anxiousness from wearing a mouthpiece, mask, and/or nasal cannula. There are no additional risks associated with high oxygen/oxygen administration for less than 24 hours as long as subjects do not have any cardiac conditions, COPD or any other lung diseases.

Subjects' answers on the health questionnaire will help the medical staff decide if they can safely participate in this study; subjects are encouraged to let the study staff know if they have any concerns.

## • Risk from Mask Application:

A mask may be applied to the subject's face using an adhesive dressing or using straps. Risks associated with mask adherence include skin irritation, redness of the skin, itchiness, tingling sensation, rash, changes in skin color, and/or headache. It is expected that some people may experience feelings of claustrophobia or anxiousness from wearing a mask.

It is expected that some people may experience increased pressure around the area of the mask, this is expected to be temporary and resolve once mask is removed.

Subjects should not take part in this study if they are allergic to adhesives. Subjects' answers on the health questionnaire will help the medical staff decide if they can safely participate in this study; subjects are encouraged to let the study staff know if they have any concerns.

## • Risk from Carbon Dioxide Administration:

Risks associated with carbon dioxide administration include dizziness, shortness of breath, drowsiness, or headache. If or when this occurs, the study can be stopped.

Other anticipated adverse events that may occur, include but are not limited to: tingling, prickling sensations ("pins and needles" feeling), restlessness, sudden increase in blood pressure, sudden increase in heart rate, sweating, and/or feeling claustrophobic or anxiousness from wearing a mouthpiece and/or mask.

These anticipated adverse events are expected to be temporary.

## • Low Oxygen Concentration Risks:

Risks associated with hypoxia include dizziness, shortness of breath, drowsiness, and/or headache. If or when this occurs, the study can be stopped.

There is an extremely small risk of loss of consciousness or death from lack of oxygen. The study shall be stopped by the subject or clinical staff long before this could occur. Breathing a hypoxic (reduced oxygen) mixture has potential risks that include damage to vital organs such as the brain, liver, kidney, and/or heart.

Other anticipated adverse events that may occur, include but are not limited to: vasovagal syncope (fainting), lightheadedness, chest discomfort (e.g. chest tightness, chest pain), feeling flush/warm, feeling of anxiety, feeling nauseated, throwing up, seizures, sudden drop in blood pressure/sudden increase in blood pressure, sudden drop in heart rate/sudden increase in heart rate, tingling sensation of face, arms and/or legs, sweating, mouth dryness, feeling claustrophobic or anxiousness from wearing a mouthpiece and/or mask. These anticipated adverse events are expected to be temporary.



Revision:

Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation

Revision:



## Nose Clip Risks:

It is expected that some people will have discomfort/pinching/scratches and/or experience symptoms similar to a headache from wearing a nose clip. If this occurs, adjustments can be made and/or the study can be stopped. The nose clip may also leave temporary indentations; these should go away shortly after the nose clip is removed.

## • Lidocaine (injection) Risks:

Injection of the Lidocaine may be discomforting and can feel like a slight pinch along with a warm/burning sensation.

Other anticipated adverse events that may occur, include but are not limited to: flushing or redness of the skin, itching skin, small red or purple spots on the skin, unusually warm skin, bruising, bleeding at the application site, swelling, feeling nauseated, dizziness, low blood pressure, and/or tremors.

Although not common, it is also possible to have an allergic reaction to injectable lidocaine (e.g., seizures). Subjects should not take part in this study if they are allergic to lidocaine injection or other types of numbing medicine, or if they have a heart rhythm disorder such as Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome. Subjects are instructed to tell the study staff right away if they experience hives; difficulty breathing; swelling of the face, lips, tongue, or throat.

These adverse events are expected to be temporary.

## • Skin Refrigerant (e.g. Ethyl Chloride, Pain Ease) Risks:

Ethyl Chloride and Pain Ease are topical anesthetics used to prevent pain by cooling the skin.

Although unlikely, the anticipated adverse events that may occur, include but are not limited to: changes in skin color (e.g., flushing or redness of the skin), delayed wound healing, rash, itching and swelling. These adverse events are expected to be temporary.

## Risk from Inflicted Knowledge:

The risk of inflicted medical knowledge to subjects is negligible since we deidentify all associated sample information including those relevant to clinical and engineering parameter studies. The monitoring and test results are not examined for diagnostic purposes and do not reflect an attempt to ascertain any subject's medical condition. The attending physician's role during this study is to ensure the safety of the subject during the study.

We will reduce the risk of inflicted knowledge by assuring the subjects that device readings and blood measurements are for research use only. In the case that a subject becomes aware of a condition (e.g., anemia, hypertension, arrhythmia etc.) they have during the study the study staff will recommend that they contact their primary care physician, and we will document this recommendation. As part of that process, we will follow up with these individuals prior to enrollment if their condition meets exclusion criteria for the study.

## • Risk From Loss of Confidentiality:

Masimo upholds the highest standards to protect hard and electronic data, however, a complete promise for confidentiality cannot be guaranteed due to unforeseeable events.

## • Risk From Additional Testing:





Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation

During the conduct of the study, it is possible, but not likely, that someone could become exposed to the sample of blood drawn from the subject through an inadvertent needle stick or by contact with an open cut. In such circumstances, it will be important to the exposed individual to know whether the blood to which he or she was exposed contained Hepatitis B Virus (HBV), Human Immunodeficiency Virus (HIV), or Hepatitis C Virus (HCV) and additional testing of the sample will be performed.

Within the consent, subjects will agree to permit a company to test the blood sample(s) by signing the consent. The test results will be maintained as confidential and will only be used by healthcare professionals for the diagnosis and treatment of the exposed individual as appropriate.

In the case that Masimo needs to contact a subject regarding additional testing, they will be contacted by a Masimo employee and medical personnel can be available for further counsel if requested.

The cost for the initial testing and compensation for their time/travel to the testing facility will be the only things paid for by Masimo.

## 4.3. Measures Taken to Protect the Rights and Welfare of Subjects

All subjects will be monitored closely throughout the study. There will be an ACLS certified medical doctor present in the study area throughout the study.

The following measures will be taken to ensure the confidentiality of the subjects:

- A code (identification) number for each subject will be kept on file.
- Only their corresponding identification number will identify subjects.
- Access to identifying documents and data will only be made to the principal investigators in the study and study staff.
- The confidentiality and retention of these documents will be protected to the extent provided and required by the law.

## 4.4. Emergency Response Plan for Medical Emergencies

The physician and nurse present during the study will be ACLS certified and will respond to any medical emergency involving a subject with the ACLS approved protocol for intervention. A crash cart equipped with medications to provide immediate care during emergencies is on site and full emergency services are within 3 miles.

## 5. OBJECTIVES OF THE CLINICAL INVESTIGATION

The primary objective of this study is to evaluate the noninvasive oxygen saturation (SpO2) performance of the noninvasive Masimo MightySat against reference arterial blood samples analyzed by a laboratory CO-oximeter reference instrument. The study will include different subgroups to assess the performance across different genders and skin pigmentation.

Data using the noninvasive devices will be collected from generally healthy male and female volunteers undergoing a desaturation procedure. Study subjects of differing levels of skin pigmentation will be enrolled in the study.

This is a nonrandomized single arm study wherein all subjects are enrolled into the experimental arm and receive the MightySat on one or more fingers. Desaturation will be conducted by reducing the concentration of oxygen the study subject breathes in a controlled manner to obtain noninvasive oxygen saturation readings, SpO2, at various levels. Reference blood samples will be repeatedly collected from the subject and analyzed using a standard laboratory CO-oximeter. The performance will be calculated using Accuracy root mean square (ARMS) analysis of the SpO2 values and the reference CO-oximeter values. An optional secondary objective of this study may be to evaluate other pulse oximetry sensors for research purposes. These sensors may include other FDA-cleared devices and commercially available pulse oximeters.

### Outcome Measure:

Performance will be determined by calculating the ARMS value through the comparison of the noninvasive oxygen saturation measurement (SpO2) to the arterial oxygen saturation (SaO2) value obtained from a reference blood sample.





Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin **Pigmentation** 

#### DESIGN OF THE CLINICAL INVESTIGATION 6.

#### 6.1. General

#### 6.1.1. **Clinical Investigation Design**

This is a nonrandomized single arm study wherein all subjects are enrolled into the experimental arm and receive the MightySat on one or more fingers. Desaturation will be conducted by reducing the concentration of oxygen the study subject breathes in a controlled manner to obtain noninvasive oxygen saturation readings, SpO2, at various levels. Reference blood samples will be repeatedly collected from the subject and analyzed using a standard laboratory CO-oximeter. The performance will be calculated using Accuracy root mean square (ARMS) analysis of the SpO2 values and the reference SaO2 values from a CO-oximeter.

#### 6.1.2. Measures Taken to Minimize/Avoid Bias:

Subjects are selected from the population surrounding the clinical research site. Where applicable, subjects with required demographics (e.g., skin pigmentation, gender, etc.) may be preferentially recruited.

#### 6.1.3. **Equipment and Materials**

Equipment and Materials: All lab analyzers and equipment will be maintained per manufacturer specifications and all study personnel will be trained on the use of relevant equipment. Equivalent equipment and materials to those listed below may be used.

## Safety Equipment (FDA-Cleared)

- Blood pressure monitoring system
- A-line pressure transducer
- Electrocardiogram (ECG)
- Masimo Pulse Oximeters (Radical-7)
- Masimo Patient Monitoring Platform (Root®)
- Pulse oximeter sensors and cables (Masimo SET, Masimo rainbow, or comparable)
- Medical-grade oxygen tank, mask, and nasal cannula
- Crash cart

## Test Devices

- Masimo MightySat investigational
- Optional: other FDA-cleared or commercially available pulse oximetry sensors



## Laboratory co-oximeters/blood analyzers

#### 6.1.4. Completion of the Clinical Investigation

The clinical investigation is considered complete when adequate data has been collected as per the sampling plan.

#### 6.2. Investigational device(s) and comparator(s)

The investigational MightySat used in this study is similar to commercially available MightySat devices

The investigational





# Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation

MightySat is equivalent to the FDA cleared version with regard to intended use on the surface of the skin, the choice of materials, biocompatibility, manufacturing process, and risk of exposure to any energy or light source. It does not pose any additional risk to patients as compared to the FDA cleared version.

Other FDA-cleared or other commercially available pulse oximeters may be used for research purposes.

## 6.3. Subjects

## 6.3.1. Eligibility Criteria

Potential subjects may be recruited and enrolled according to the criteria below.

## **Inclusion Criteria (Eligible Subjects)**

- Subject is 18 to 50 years of age.
- Subject weighs a minimum of 110 lbs.
- Subject has a hemoglobin value  $\geq 11$  g/dL.
- Subject's baseline heart rate is  $\geq 45$  bpm and  $\leq 85$  bpm.
- Subject's CO value is  $\leq 2.0\%$  FCOHb.
- Subject's blood pressure: Systolic BP ≤ 140 mmHg and ≥ 90 mmHg, Diastolic BP ≤ 90 mmHg and ≥ 50 mmHg, and if systolic BP is lower than 100 mmHg and/or diastolic BP is lower than 60 mmHg, subject passes an orthostatic blood pressure test.
- Subject is able to read and communicate in English and understands the study and the risks involved.

## Exclusion Criteria (Ineligible Subjects) (\* = Per Physician Discretion)

- Subject is pregnant.
- Subject has a BMI > 35.
- Subject has a history of fainting (vasovagal syncope), blacking out or losing consciousness during or after a blood draw, or has a fear of blood draws.
- Subject has open wounds, inflamed tattoos or piercings, and/or has any visible healing wounds that a medical professional determines may place them at an increased risk for participation.\*
- Subject has known drug or alcohol abuse.
- Subject uses recreational drugs.\*
- Subject experiences frequent or severe headaches and/or migraine headaches, migraine auras, altitude sickness, and/or headaches accompanied by visual changes or sensitivity to light or sound.
- Subject has experienced a concussion or head injury with loss of consciousness within the past 12 months.
- Subject has any history of a stroke, myocardial infarction (heart attack), and/or seizures.
- Subject has any chronic bleeding disorder (e.g. hemophilia).
- Subject has taken anticoagulant medication within the past 30 days (excluding nonsteroidal antiinflammatory drugs (NSAIDS)).
- Subject has donated blood within the past 4 weeks.
- Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome.
- Subject has any symptomatic cardiac dysrhythmia (e.g. atrial fibrillation) and has not received clearance from their physician to participate.
- Subject has a known neurological and/or psychiatric disorder (e.g. schizophrenia, bipolar disorder, multiple sclerosis, Huntington's disease) that interferes with the subject's level of consciousness.\*
- Subject has taken opioid pain medication 24 hours before the study.
- Subject has any active signs and/or symptoms of infectious disease (e.g. hepatitis, HIV, tuberculosis, flu, malaria, measles, etc.).\*
- Subject is taking medications known to treat any type of infectious disease.
- Subject has either signs or history of peripheral ischemia or carpal tunnel syndrome.
- Subject has had invasive surgery within the past year, including but not limited to major dental surgery, appendectomy, plastic surgery, jaw surgery, major ENT surgery, major abdominal and/or pelvic surgery, heart surgery, or thoracic surgery.\*
- Subject has symptoms of congestion, head cold, or other illnesses.





## Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin **Pigmentation**

- Subject has been in a severe car accident(s) or a similar type of accident(s) requiring hospitalization within the past 12 months.
- Subject has any cancer or history of cancer (not including skin cancer).\*
- Subject has chronic unresolved asthma, lung disease (including COPD) and/or respiratory disease.
- Subject is allergic to lidocaine, chlorhexidine, latex, adhesives, or plastic.
- Subject has a heart condition, insulin-dependent diabetes, or uncontrolled hypertension.
- Subject has delivered vaginally, has had a pregnancy terminated, a miscarriage with hospitalization, or had a C-section within the past 6 months.
- Subject intends on participating in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle, tennis), exercise (working out, riding a bike, riding a skateboard, etc.), or any activity that will put additional stress on the wrist within 24 hours following a study that involves an arterial line.
- Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of the investigator/study staff.

#### 6.3.2. **Expected Duration of the Clinical Investigation and Subject Participation**

Expected duration of study enrollment is 3 to 6 months.

Subject participation in the study will be approximately 180 minutes.

#### 6.3.3. Withdrawal of Subjects

Subjects must be withdrawn under the following circumstances: the subject withdraws consent, or at the discretion of investigator/study staff for subject safety and welfare.

#### 6.3.4. Replacement of Subjects

In case a subject is withdrawn from the study, another subject may be recruited.

#### 6.3.5. **Re-contacting Subjects**

If the subject fails to provide proper documentation on their individual consent form or other study documents, Masimo may re-contact the subject and ask them to return to the clinical lab in order to properly complete these documents. The subject will be re-contacted via phone or email and be asked to return as soon as possible. The subject will be compensated for travel.

#### 6.3.6. **Vulnerable Populations**



The study may also enroll subjects who are economically disadvantaged, unemployed and/or educationally disadvantaged. Reasonable compensation will be provided for economically disadvantaged subjects to eliminate possibility of undue influence due to financial incentive. Educationally disadvantaged subjects will be provided ample time to ask questions and comprehend information.

#### 6.4. **Procedures**







Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation



## 6.4.2. Recruitment and Prescreening

Subjects will be recruited using IRB-approved advertisements. Subjects may be referred to the study by previous subjects. Subjects are contacted via phone call to conduct a prescreening interview to determine their initial eligibility for the study. Potential eligible subjects are scheduled for a study visit to the clinical laboratory.

## 6.4.3. Consenting and Screening

Subjects will be asked to provide a copy of their valid government-issued identification such as driver's license and/or Social Security card. Copies of these forms of identification will be stored electronically. Subjects must read and sign the IRB-approved informed consent document. No study related activities will be conducted until the consent form is signed.

After informed consent is obtained, subjects will be asked a brief series of health questions to ensure their eligibility for this study. Subjects who do not meet the inclusion criteria and/or meet exclusion criteria will not be eligible to participate in the study.

Subject demographic information including age, sex, pigmentation, ethnicity, height and weight will be collected. These may be recorded for data analysis and/or subject safety monitoring purposes.





Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation

The objectives of this study require subjects with a range of skin pigmentations to be enrolled.

Therefore, all subjects will need to undergo a skin pigmentation screening to maintain sample size requirements.

Body mass index (BMI) may also be calculated to assess for eligibility for the study.

In addition, a medical history will be recorded after the initial screening questionnaire. Vital signs, such as blood pressure and heart rate, will be recorded for subject safety monitoring. Pulse oximetry measurements, such as SpO2, SpCO, and SpHb, may also be recorded.

An orthostatic blood pressure test is ONLY required to be performed on subjects that meet the following criteria:

- Initial systolic blood pressure lower than 100 mmHg and greater than or equal to 90 mmHg, and/or
- Initial diastolic blood pressure lower than 60 mmHg and greater than or equal to 50 mmHg.

The following combinations meet the criteria for performing an orthostatic blood pressure measurement. If the criteria are not met, an orthostatic blood pressure test is not required.

Table 1: Criteria for orthostatic blood pressure measurement.

| Systolic measurement (mmHg) | Diastolic measurement (mmHg) | Perform orthostatic blood pressure test? |
|---|---|---|
| 100 or above | 50 to 59 | YES |
| 90 to 99 | 60 or above | YES |
| 90 to 99 | 50 to 59 | YES |
| 100 or above | 60 or above | NO |

The orthostatic blood pressure test will start with the clinician taking the subject's blood pressure while they are lying in supine position. The subject will then stand up for 30 seconds and a second blood pressure measurement will be taken. The subject's blood pressure will need to stay above 90/50 to meet inclusion criteria for the study.

Female subjects will be required to take a pregnancy test. Results will be noted in study documentation. If the pregnancy test is positive, the subject will be notified and removed from the study.

A venous sample will be obtained via needle stick or by placement of an IV and analyzed to verify that the starting hemoglobin level is greater than or equal to 11 g/dL and carboxyhemoglobin (COHb) level is less than or equal to 2.0%. If hemoglobin level is less than 11 g/dL and/or COHb is greater than 2.0%, the subject will be excluded from the study.

### 6.4.4. Procedure

The subject will be seated and/or lying-in supine position and should refrain from excessive movement during the study.

If accepted into the study, the subject's vitals will be monitored with standard noninvasive monitors, including FDA-cleared pulse oximeters, ECG, and blood pressure cuff. Information from these monitors may optionally be recorded.

Transient increases in blood pressure and heart rate can be expected during line placement, needle sticks, blood draws etc. and may also be attributed to anxiety/nervousness relating to a new environment. For most participants, only the initial recorded blood pressure and/or heart rate determines a subject's qualification for the study. In the case where heart rate and blood pressure





Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation

changes suggest participant discomfort or a potential safety concern, the participant will be removed from the study after qualifying, according to the discretion of medical and study staff.

A peripheral venous line will be placed in the subject's hand or arm. This line may be used for the qualifying venous blood draw and for safety or clinical intervention required during the study. The peripheral venous line site will be observed by study staff prior to line placement to ensure no bruising remains from any previous IV placements; if there is bruising the clinician will place the line in another location.

Local anesthetics such as lidocaine or skin refrigerant (e.g. Ethyl Chloride or Pain Ease) may be used if an IV is placed, to numb the site. Subjects will be given the option to have lidocaine or numbing spray be used during IV placement for the purpose of making catheter placement more comfortable.

After intravenous access is established, one or more intra-arterial catheter(s) (arterial line or A-line) will be placed in the radial artery of the subject's wrist. Lidocaine will be used to ease discomfort. This study will be done with an arterial line to facilitate continuous blood pressure measurement, and to allow for blood sampling from this site to determine arterial blood gas values (ABG) such as oxygen saturation. Noninvasive ultrasound devices may be used to facilitate line placement.

Upon successful placement of the IV(s), arterial line(s) and the subject's indication that they are comfortable, a minimum of one FDA-cleared pulse oximeter sensor will be placed on the subject for reference values such as oxygen saturation.

After arterial access is established, the study sensor(s) will be placed on the subject's finger(s). Data collection will be initiated . Sensors may be repositioned, as needed, to ensure proper placement.

Pulse oximeter output values (e.g., SpO2, pulse rate) will be recorded using the data collection software. Raw absorbance data from the noninvasive device(s) will also be recorded using the data collection software.

Upon successful placement of the sensors and the subject's indication that they are comfortable, a baseline set of blood samples will be obtained.

A qualified person will complete blood draws. Arterial blood samples may be drawn consecutively during the procedure at different saturation levels. No more than 100 samples of approximately 1-4 cc each may be drawn including blood drawn to flush the line and prepare for new samples. A maximum total of 275 cc of blood may be taken per subject.

Subjects may wear a nose clip or nose plugs and use a mouthpiece, or wear a mask, during the desaturation procedure. The mask may be secured to the subject's face by securing adjustable straps and/or Tegaderm adhesive (or equivalent) to secure mask to skin. Subjects may be asked to shave the area of application to allow the mask to stick to skin. The area of application may also be wiped to remove facial oils, make-up, or any other skin products. End-tidal and/or partial pressure of carbon dioxide and respiration rate values will be noted at the beginning of the desaturation portion of the study for subject safety purposes and will be noted again at the end of the desaturation portion of the study. If respiratory rate is greater than 30 breaths per minute at room air (21% FiO2), the study will be stopped. If respiratory rate is less than or equal to 5 breaths per minute at room air (21% FiO2), check blood gas values of first samples after the mouthpiece or mask is placed, then the study will proceed.

Upon indication that the subject is comfortable, a gas mixture will be administered through the mouthpiece. The gas mixture may include varying proportions of oxygen, carbon dioxide, and nitrogen. The proportion of oxygen in this mixture will be decreased in a controlled manner to lower the subject's blood oxygen saturation. The lowest targeted value will be 70% oxygen saturation. Readings near 70% will be immediately verified by the reference CO-oximeter to ensure that levels are





Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation

within the targeted oxygen saturation range and to minimize time that the subject may drop below the targeted range. At any point in the study, if the subject feels uncomfortable, the subject will be given oxygen.

Subjects may undergo the desaturation procedure up to 3 times.



after the procedures. If at any point the subject is uncomfortable with the study, the study will be stopped.

Oxygen tank pressure will be checked and noted before the study begins for subject safety purposes.

During the study, subjects may be recorded using photography and/or videography. The recordings may include sound. These recordings may capture identifying features on the hand and/or arm. These recordings may be used in research, product development, product testing, training, and comparison study purposes. Subjects will be given the option to provide consent or opt-out of the recordings

## 6.4.5. Ending Procedure

Study staff may take one final blood draw of 1-4cc, in addition to the blood draws in the procedure section above, to verify the subject's blood values are within normal ranges (e.g., pH, glucose, etc.).

The total overall lab time will be approximately 180 minutes. In the event that the total lab time exceeds 180 minutes, subjects will be compensated for the extra time. Subjects will be paid according to the compensation breakdown on the consent form.

At the conclusion of the procedure, the sensor(s)/device(s), IV(s), and arterial line(s) will be removed. A set of pre-discharge vitals, such as heart rate and blood pressure, will be obtained and recorded on the case report form for subject safety purposes. Subjects will be given instructions on post care. All subjects will be instructed to contact the principal investigator or study staff in the event of any potential complication.

Subjects will be offered a snack and water or juice. Subjects are asked to consume food and/or liquid prior to leaving the clinical lab area for their safety due to study procedures such as blood removal and line placement. Subjects may also be asked to wait in the clinical lab or lobby waiting area for up to an additional 30 minutes before leaving to allow for their body to continue adjusting after the study has completed.

All subjects will be encouraged to remain in the study area until they feel fit to leave. Subjects should feel safe and able before returning to work directly after participation in the study. All subjects, will be advised to take as much time as they need after the study before returning to work.

The subject will be allowed to leave after medical personnel determine it is safe to do so.

## 6.5. Monitoring plan

A separate document for the study monitoring plan will be developed and followed to ensure subject safety and GCP compliance.

## 7. STATISTICAL DESIGN AND ANALYSIS

## 7.1. Acceptance Criteria

For validation studies, acceptance criteria are determined by Masimo specifications for each design.

### 7.2. Sample Size



Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation



- d. The final  $A_{RMS}$  analysis will utilize statistical methods to ensure performance statistics are calculated with comparable density over the range 70-100% SaO<sub>2</sub> and account for multiple samples per subject.
- e. Statistical analysis for each subgroup will be performed to show differences in biases among different subgroups.
- f. Depending on dropout rates, additional subjects may be enrolled to obtain sufficient representative data for factors such as gender, skin pigmentation, oxygen saturation, and other factors as required.

## 7.3. Statistical Analysis

a. Exclusion

The following data exclusion criteria will be applied before statistical analysis:

- i. Either reference or test device does not provide data;
- ii. Incomplete study or early termination, where the desaturation protocol could not be completed;
- iii. Reference device malfunctions and/or provides inconsistent saturation values;
- iv. Discontinuities and abrupt dropouts due to instruments recalibration or device failure;
- v. Low signal quality, e.g. due to noise or interference.



- vii. Exclusion of subjects that do not have desaturation points in the lowest saturation bin.
- viii. Exclusion of data to statistically equalize samples per subject, and across the 70-100% saturation bins.
- b. Accuracy calculations

Accuracy will be reported as the Bias, Precision and A<sub>RMS</sub> using the following equations:

$$Bias = \frac{1}{n} \sum_{i=1}^{n} (SpO2 - SaO2)$$

$$Precision = \sqrt{\frac{\sum_{i=1}^{n} ((SpO2 - SaO2) - Bias)^{2}}{n}}$$





Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin **Pigmentation** 

**Revision:** 

$$A_{RMS} = \sqrt{\frac{\sum_{i=1}^{n} (Sp02 - Sa02)^{2}}{n}}$$

The A<sub>RMS</sub> and precision values will be adjusted to account for repeated measurements on each subject.

#### 7.4. **Expected Dropout Rates**

Subjects may not complete the study for various reasons, such as screen failure, they are unable to complete desaturation criteria, or they are unable to have intravenous or arterial line placed. Expected drop out rate for this study is approximately 50% of the subjects who consented to participation in this study.

#### 8. **DATA MANAGEMENT**

#### 8.1. Data Management and Confidentiality

All documents associated with this protocol will be securely stored in a physical location or on password-protected computers. The confidentiality and retention of these documents will be protected to the extent provided and required by the law. All data will be de-identified before any statistical analysis. Only de-identified data will be shared with Masimo for research purposes stated in this protocol. Data collected by data capture software and data entered in case report form will be shared with Masimo via a secure, password-protected server that only study staff and Masimo study team members will have access to. Data will be retained for a minimum to 2 years following completion of the final analysis.

#### 8.2. **Source Documents**

Source data is all information, original records of clinical findings, observations, or other activities in a clinical trial necessary for the reconstruction and evaluation of the trial. Source data are contained in source documents. Examples of these original documents and data records include: hospital records, clinical and office charts, laboratory notes, memoranda, recorded data from automated instruments, and copies or transcriptions certified after verification as being accurate and complete.

#### 8.3. Case Report Forms

The site shall capture study data in case report forms (CRFs) for each subject enrolled, to be provided to the sponsor. CRFs may be in paper or electronic format through electronic data capture (EDC) software. Masimo shall ensure that systems used for electronic CRFs are compliant with the requirements of 21 CFR Part 11 and ISO / IEC 27001 Certification. The CRFs will be completed and signed by the principal investigator or delegate. This also applies to those subjects who fail to complete the study. If a subject withdraws from the study, the reason must be noted on the CRF. Case report forms are to be completed on an ongoing basis. CRF entries and corrections will only be performed by study site staff, authorized by the investigator. For paper CRFs, entries and corrections to the CRF will be made following Good Documentation Practices.

The CRF may include the following information, including but not limited to: inclusion / exclusion criteria, whether subject consent was obtained before start of study, demographic information, device readings, and if occurrence of any adverse event, protocol deviation, and device deficiencies, etc. The CRFs will be signed by the PI or delegate to attest that the data are complete and accurate.

CRF entries will be checked by the study monitor and any errors or inconsistencies will be queried to the site on an ongoing basis. Any changes made within an electronic CRF will be tracked by audit trail. Any changes on a paper CRF will be made directly on the CRF and will be initialed and dated by the person making the change. Query resolution will be assessed and confirmed by study monitor during site visit.

#### 8.4. **Data Transfer and Storage**

- Original paper CRFs will be stored in a secure location at the site. Copy of the original paper CRFs may be scanned and sent to sponsor. If using electronic CRFs, the site staff will be assigned unique usernames and passwords for data security. Final copies of the electronic CRFs in EDC are stored on a secure server.
- 8.4.2. Only authorized sponsor personnel will have access to study data, and will move it to a secure and backed-up drive at Masimo.
- CRFs will be checked for completeness and if there are inconsistent or missing data points, queries will be 8.4.3. generated. If delegated study staff are to correct the paper CRF, they shall follow GDP practices to strike





Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation

through old entry, add in new entry, and initial and date it, and provide the corrected information to sponsor. Corrections made to electronic CRFs will be tracked by audit trail and require PI or delegate sign-off.

## 8.5. Record Retention

Study data will be retained for the necessary period of time as required by the institution's regulations. Study records shall be retained for a minimum of two years after study closure. The Institution's own retention policies and regulations may apply in addition to the minimal requirement.

## 9. AMENDMENTS TO THE CLINICAL INVESTIGATION PLAN

Any changes made to the clinical investigational plan/study protocol will be documented by way of an amendment. Before submitting a protocol amendment to the IRB, the protocol amendment must be agreed upon and signed by both the principal investigator and the sponsor. The protocol amendment will be submitted to the IRB for approval. At a minimum, a redline version and a clean version of the new protocol amendment will be kept on file by the PI and the sponsor. Protocol amendments will need to be version controlled. Both PI and sponsor will retain the IRB approval letter as confirmation that the protocol amendment was approved.

## 10. DEVIATIONS FROM CLINICAL INVESTIGATION PLAN

Deviations from the protocol must receive both Sponsor and the investigator's IRB/ethics committee approval before they are initiated, with the exception that under emergency circumstances, deviations from the Clinical Investigation Plan to protect the rights, safety and well-being of human subjects may proceed without prior approval of the sponsor or the IRB/ethics committee. Any protocol deviations initiated without Sponsor and the investigator's IRB/ethics committee approval that may affect the scientific soundness of the study, or affect the rights, safety, or welfare of study subjects, must be documented and reported to the Sponsor and to the investigator's IRB/ethics committee as soon as a possible, but no later than 5 working days after the occurrence of the protocol deviation. In addition to documenting deviations on the CRF, the Protocol Deviation Form may also be used. If protocol deviations continue to occur frequently at a study site, a corrective and preventive action (CAPA) may be opened by the Sponsor.

**Withdrawal of IRB approval:** An investigator shall report to the sponsor a withdrawal of approval by the investigator's reviewing IRB as soon as possible, but no later than 5 working days of the IRB notification of withdrawal of approval.

## 11. DEVICE ACCOUNTABILITY

## 11.1. Receipt of Study Device

Upon receipt of the of the study device supplies, an inventory must be performed and the device accountability log filled out and signed by the person accepting the shipment. It is important that the designated study staff counts and verifies that the shipment contains all the items noted in the shipment inventory. Any damaged or unusable study devices in a given shipment will be documented in the study files. The investigator must notify the study sponsor of any damaged or unusable study devices that were supplied to the investigator's site.

## 11.2. Use of Study Device

Use of study device will be documented on case report forms for each subject. Any unused devices must be returned to the Sponsor at the end of the study or before product expiration date.

## 11.3. Return or Destruction of Study Device

At the completion of the study, there will be a final reconciliation of study devices shipped, devices used, and devices remaining. This reconciliation will be logged on the device accountability log. Any discrepancies noted will be investigated, resolved, and documented prior to return or destruction of unused study devices. Devices destroyed on site will only be upon written instruction from the sponsor and will be documented in the study files. When a Masimo device deficiency is observed, every effort should be made to return the device and its packaging to the Sponsor in a timely manner.

## 12. STATEMENTS OF COMPLIANCE

This document is a clinical investigational plan for a human research study sponsored by Masimo Corporation. The study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki. By participating in the study, the Investigator agrees to adhere to all stipulations of this protocol, the conditions of the Institutional Review Board (IRB)





# Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation

or Research Ethics Committee approval, federal and local regulatory requirements, 21 CFR 812, ISO-14155, International Conference on Harmonization Good Clinical Practice (ICH GCP) guidance.

The protocol, informed consent form(s), recruitment materials, and all participant materials will be submitted to the Institutional Review Board (IRB) for review and approval. Approval of both the protocol and the consent form must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study.

### 13. INFORMED CONSENT PROCESS

Subjects must read and sign the consent document using the informed consent process as outlined in FRM-3451 Informed Consent Process. No study-related activities will take place prior to informed consent.

## 14. ADVERSE EVENTS, ADVERSE DEVICE EFFECTS, AND DEVICE DEFICIENCIES

### 14.1. Definitions

The definitions for adverse event, adverse device effect, serious adverse event, serious health threat, serious adverse device effect, and unanticipated adverse device effect, device deficiencies are provided below (ISO 14155, 21 CFR 812.3(s)).

- <u>adverse event</u>: untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device and whether anticipated or unanticipated (ISO 14155)
- adverse device effect: adverse event related to the use of an investigational medical device
- <u>serious adverse event</u>: adverse event that led to any of the following:
  - o a) death
  - o b) serious deterioration in the health of the subject, users, or other persons as defined by one or more of the following:
    - 1) a life-threatening illness or injury, or
    - 2) a permanent impairment of a body structure or a body function including chronic diseases, or
    - 3) in-patient or prolonged hospitalization, or
    - 4) medical or surgical intervention to prevent life-threatening illness or injury, or permanent impairment to a body structure or a body function,
  - o c) fetal distress, fetal death, a congenital abnormality, or birth defect including physical or mental impairment

Note: Planned hospitalization for a pre-existing condition, or a procedure required by the Clinical Investigation Plan, without serious deterioration in health, is not considered a serious adverse event.

- <u>serious health threat</u>: signal from any adverse event or device deficiency that indicates an imminent risk of death or a serious deterioration in the health in subjects, users or other persons, and that requires prompt remedial action for other subjects, users or other persons.
  - Note: This would include events that are of significant and unexpected nature such that they become alarming as a potential serious health hazard or possibility of multiple deaths occurring at short intervals.
- <u>serious adverse device effect</u>: adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event
- <u>unanticipated serious adverse device effect</u>: serious adverse device effect which by its nature, incidence, severity or outcome has not been identified in the current risk assessment
  - Note: Anticipated serious adverse device effect (ASADE) is an effect which by its nature, incidence, severity or outcome has been identified in the risk assessment.
- <u>device deficiency</u>: inadequacy of a medical device with respect to its identity, quality, durability, reliability, usability, safety or performance





# Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation

Note 1: Device deficiencies include malfunctions, use errors, and inadequacy in the information supplied by the manufacturer including labelling.

Note 2: This definition includes device deficiencies related to the investigational medical device or the comparator.

## 14.2. List of non-reportable adverse events

All adverse events will be reported to Sponsor.

## 14.3. Adverse Event Reporting

- All Adverse Events, both Anticipated and Unanticipated, must be recorded in the CRF and in the Adverse Event Report Form.
- All Adverse Events must be promptly reported to the Sponsor.
- All Unanticipated Adverse Device Effects will be also reported to both the Sponsor and the IRB.
- Both Serious Adverse Events and Unanticipated Adverse Device Effects must be reported to the Sponsor within 48 hours. All other Adverse Events should be reported to the Sponsor within 5 business days.
- All Serious Adverse Events will be also reported to the IRB per IRB reporting requirements. These reports may include, but will not be limited to: date of onset; brief description of the events; their treatment; whether they resulted in death, inpatient hospitalization, severe or permanent disability or were life threatening; their relationship to the study device; and resolution.

## 14.4. Device Deficiencies Reporting

All Masimo device related deficiencies should be reported to the Sponsor and must be recorded in the CRF in a timely manner. When a Masimo device deficiency is observed, every effort should be made to return the device and its packaging to the Sponsor in a timely manner. Vulnerable population

### 14.5. Definition

Vulnerable population are research participants, such as children, prisoners, pregnant women, handicapped, or mentally disable persons, or economically or educationally disadvantaged persons, who are likely to be vulnerable to coercion and undue influence.

The federal regulations that govern the protection of human subjects require additional protection for the vulnerable population.

## 14.6. Protection of vulnerable subjects



- Reasonable compensation will be provided for economically disadvantaged subjects to eliminate possibility of undue influence due to financial incentive.
- Educationally disadvantaged subjects will be provided ample time to ask questions and comprehend information.
- Medical care will be provided to these subjects after the clinical investigation has been completed if they are injured as a
  direct result of participating in this research study. The cost of treatment for any research related injury will be covered
  by Masimo.

## 14.7. Responsible Parties

- The IRB will review research with vulnerable populations and evaluate consent, level of risk, coercion, and the reason for choosing this particular subject population. The IRB will be responsible for determining what practices will include continuing review for compliance while monitoring these studies.
- The Investigator holds the ultimate responsibility for protecting the rights, safety, and welfare of research subjects by ensuring that all regulations and proper documentation of consent is handled in a compliant and timely manner.





Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin **Pigmentation** 

#### 15. SUSPENSION OR PREMATURE TERMINATION OF THE CLINICAL INVESTIGATION

#### 15.1. Suspension or Termination of Study Site

The sponsor can suspend or prematurely terminate the PI's and study site's participation in the study, particularly if sponsor finds serious non-compliance by the PI or site, and if such non-compliance was not resolved in a timely manner. The sponsor will document the decision to suspend or terminate the investigation in writing. A suspended study site cannot enroll new subjects.

If the sponsor determines that the study site's compliance to be inadequate at any point during the study, and sponsor move to suspend or terminate the study site, the sponsor will provide notification in writing to the principal investigator and IRB as necessary. The study site is eligible for reinstatement upon correction of any findings and any open action items prior to the suspension along with a written guarantee that the same non-compliance will not reoccur in the future. Site can only resume subject enrollment upon receiving written notification of reinstatement from the sponsor.

If for any GCP and Regulatory non-compliance reasons the study site is prematurely terminated by the sponsor, then the study site is not eligible for reinstatement under the same Clinical Investigational Plan/Study Protocol.

#### 15.2. Termination of Clinical Investigation/Study due to UADE

The clinical investigation may be terminated if sponsor determines that an unanticipated adverse device effect presents an unreasonable risk to the subjects. Termination shall occur not later than 5 working days after the sponsor makes this determination, and not later than 15 working days after the sponsor first received notice of the effect.

The sponsor may resume the terminated clinical investigation with prior IRB approval if the device is non-significant risk.

#### 16. **PUBLICATION POLICY**

In compliance with 42 CFR Part 11, a study that meets the definition of an Applicable Clinical Trial (ACT) and that is initiated after September 27, 2007 must be registered on ClinicalTrials.gov. Results of the clinical investigation will be made publically available.

| 17. | BIBLIOGRAPHY |
|-----|--------------|

#### 18. **REVISION HISTORY**

| Version Number | Version Date | Summary of Revisions Made |
|----------------|--------------|---------------------------|